CLINICAL TRIAL: NCT05826262
Title: Role of Laparoscopy in Penetrating Anterior Abdominal Wall Injuries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Omar Ragheb, resident at general surgery department, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-23-03-16MS
Record Dates: First submitted 2023-03-20; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Evaluate Laparoscopic Management in Patients With Penetrating Anterior Abdominal Wall Trauma
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with penetrating anterior abdominal wall injuries (Experimental)
  Interventions: Procedure: diagnostic laparoscopy

INTERVENTIONS:
Procedure: diagnostic laparoscopy — diagnosis and management of patients with penetrating anterior abdominal wall injuries

SUMMARY:
The current study is aiming to evaluate the diagnostic and therapeutic role of laparoscopy in patients with penetrating anterior abdominal wall trauma as regard the accuracy of diagnosis and efficacy in management and avoidance of unnecessary laparotomy

ELIGIBILITY:
Inclusion Criteria:

* All patients with penetrating anterior abdominal wall injuries Age will be between 5 - 65 years old

Exclusion Criteria:

* Vitally unstable patients Patients with associated injuries

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-03-10 (Estimated); Study Completion 2024-03-10 (Estimated)

PRIMARY OUTCOMES:
Morbidity | 1 month

SECONDARY OUTCOMES:
Mortality | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided